CLINICAL TRIAL: NCT01357525
Title: SBRT for Close or Positive Margins After Resection of Pancreatic Adenocarcinoma A Prospective Evaluation in Select Patients With Resected Pancreas Cancer
Brief Title: SBRT for Close or Positive Margins After Resection of Pancreatic Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David A. Clump, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, David A. Clump, MD, PhD, Assistant Professor, Radiation Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 10-123
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Adenocarcinoma of the Pancreas
Keywords: Pancreas; Resected
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Stereotactic Body Radiotherapy (Other)
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — An SBRT plan will be created by a medical physicist based on the PTV contoured on the CT scan. The plan will be to deliver fractionated SBRT to the isodose line best encompassing the PTV:
  12 Gy x 3 fractions (36 Gy total)
  Other Names: CyberKnife; Trilogy; True Beam; Radiosurgery; SBRT

SUMMARY:
The current study seeks to further investigate the impact of Stereotactic Body Radiation Therapy following pancreatic resection with a close or positive margin. The investigators hope to improve local control, and through the use of a shortened treatment schedule, allow patients to begin systemic therapy earlier.

DETAILED DESCRIPTION:
Radiation simulation will be done in Shadyside Radiation Oncology department Contrast-enhanced CT based simulation will be obtained prior to any adjuvant treatment (2-4 weeks post-op depending on healing). The target volume will be identified based on fiducial marker placement at time of surgery as well as a detailed discussion and image review with the operating surgeon. This are will be contoured on axial CT images obtained at 1.25 mm slice thickness. These volumes will then be reconstructed into a 3-dimensional image set for SBRT planning. Subjects will be simulated in the treatment position (supine with arms raised) on the CT scanner table the appropriate immobilization. Optiray® contrast will be administered intravenously at a flow rate of 2.5 mL/s. A helical CT scan of the abdomen will be acquired with intravenous contrast starting 30 seconds prior to CT acquisition.

A 4D CT data acquisition for the same axial extent will be obtained. The images will then be electronically transferred from the CT workstation via DICOM3 to the appropriate treatment planning workstation in the department of radiation oncology. Based on axial CT images, fiducial marker placement, review of the pathology report, and a detailed discussion with the operating surgeon, contours will be drawn of the clinical target volume (CTV), which is defined as the area at risk for microscopic disease. The planning target volume (PTV) will be equivalent to the CTV unless motion is detected on the 4D motion study. If there is motion, the amount of motion in the superior-inferior, lateral, and anterior-posterior directions will be the margin given. Surrounding normal and critical structures will also be contoured by the treating radiation oncologist including the kidneys, liver, small bowel, spinal cord, and stomach if necessary.

Stereotactic Body Radiotherapy Planning An SBRT plan will be created by a medical physicist based on the PTV contoured on the CT scan. The plan will be to deliver fractionated SBRT to the isodose line best encompassing the PTV.

Careful evaluation of each plan will be conducted by the radiosurgical team to ensure that normal tissues and critical structures tolerances are maintained.

The maximum dose (in Gy) within the treatment volume (MD), prescriptions dose (PD), and the ratio of MD/PD (as a measure of heterogeneity within the target volume), prescription isodose volume (PIV in mm3), tumor volume (TV in mm3), and the ratio of PIV/TV (as a measure of dose conformity of the treatment relative to the target) will be recorded.

Evaluation during treatment The subjects will be carefully followed while on active treatment and post-treatment for 24 months, or until death.

Treatment following SBRT All patients will have been seen in a multi-disciplinary pancreatic cancer clinic. As such, they will be set up with a medical oncologist. Following completion of SBRT as described in this protocol, the patient's medical oncologist may, at his/her discretion, administer systemic therapy according to the current standard of care or the UPMC pathways.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the pancreas that has been resected with a close (<2.5mm) or positive margin based on surgical and pathological findings.
* Subjects will be staged according to the 2010 AJCC staging system (Appendix E) with pathologic stage T1-4, N0-1 being eligible; and have a primary tumor of the pancreas (i.e., pancreatic head, neck, uncinate process, body/tail
* PTV must be encompassed in a reasonable SBRT "portal" as defined by the treating radiation oncologist
* Karnofsky performance status > 70 (ECOG 0-1)
* Age > 18
* Estimated life expectancy > 12 weeks
* Patient must have adequate renal function as defined by serum creatinine<1.5mg/dl obtained within 28 days prior to registration
* Patient must have adequate hepatic function as defined by total bilirubin <1.5 xIULN(institutional upper limit of normal) and either SGOT or SGPT <2.5xIULN, obtained within 28 days prior to registration.
* Patient must be able to swallow enteral medications. Patient must not require a feeding tube. Patient must not have intractable nausea or vomiting, GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, or uncontrolled inflammatory bowel disease (Chron's, ulcerative colitis).
* Ability to provide written informed consent
* Patient must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, history of myocardial infarction or cerebrovascular accident within 3 months prior to registration, uncontrolled diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not be pregnant because of the risk of harm to the fetus. Nursing women may participate only if nursing is discontinued, due to the possibility of harm to nursing infants from the treatment regimen. Women/men of reproductive potential must agree to use an effective contraception method.

Exclusion Criteria:

* Non-adenocarcinomas, adenosquamous carcinomas, islet cell carcinomas, cystadenomas, cystadenocarcinomas, carcinoid tumors, duodenal carcinomas, distal bile duct, and ampullary carcinomas are not eligible.
* Evidence of distant metastasis on upright chest x-ray (CXR), computed tomography (CT) or other staging studies
* Subjects with recurrent disease
* Prior radiation therapy to the upper abdomen or liver
* Prior chemotherapy
* Subjects in their reproductive age group should use an effective method of birth control. Subjects who are breast-feeding, or have a positive pregnancy test will be excluded from the study
* Any co-morbidity or condition of sufficient severity to limit full compliance with the protocol per assessment by the investigator
* Concurrent serious infection
* Previous or current malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in situ, adequately treated basal cell or squamous cell carcinoma of the skin, and treated low-risk prostate cancer.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02-06 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Clump, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Body Radiotherapy
Started | 50
Completed (Participant underwent surgery but did not receive SBRT.) | 49
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Patients that received treatment.
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 69.9 [62.2 to 75.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Local Progression-free Survival (LPFS) at 1-year
Description: Percentage of patients that did not experience progressive disease (PD) in the target lesion. Death or development of distant disease was not regarded as an event. For patients that underwent surgical resection, local progression was defined as disease recurrence detected on follow-up imaging (CT or FDG-PET/CT) that is located within the SBRT target volume.
Time Frame: Up to 12 months
Population: Patients that received study treatment per protocol and were evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 43
percentage of participants | 85

2. Primary Outcome: Local Progression-free Survival (LPFS) at 2-years
Description: as for outcome 1
Time Frame: Up to 24 months
Population: Patients that received study treatment per protocol and were evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 43
percentage of participants | 78.12 [57.82 to 93.06]

3. Primary Outcome: Local Progression-free Survival (LPFS)
Description: Percentage of patients without disease progression in target lesion from time from enrollment until one month. Death or development of distant disease is not regarded as an event. For patients that undergo surgical resection, local progression will be defined as disease recurrence detected on follow-up imaging (CT or FDG-PET/CT) that is located within the SBRT target volume.
Time Frame: Up to 24 months
Population: Patients that received study treatment per protocol and were evaluable for response.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 49
percentage of participants | NA [41 to NA] — Median not determined; upper bound not reached

4. Primary Outcome: Regional Progression-free Survival (RPFS)
Description: Time duration that patients that did not experience progressive disease (PD) in the target lesion. Death or development of distant disease was not regarded as an event. For patients that underwent surgical resection, local progression was defined as disease recurrence detected on follow-up imaging (CT or FDG-PET/CT) that is located within the SBRT target volume.
Time Frame: Up to 24 months
Population: Patients that received study treatment per protocol and were evaluable for response.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 49
months | NA [27 to NA] — Median not determined; Upper bound not reached.

5. Primary Outcome: Regional Progression-free Survival (RPFS) at 2-years
Description: as for outcome 1
Time Frame: Up to 24 months
Population: Patients that received study treatment per protocol and were evaluable for response.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 49
percentage of participants | 72.2 [57.56 to 87.84]

6. Primary Outcome: Distant Metastasis-free Survival (DMFS) at 2 Years
Description: Percentage of patients that did not experience distant metastasis. Death or development of distant disease was not regarded as an event. For patients that underwent surgical resection, local progression was defined as disease recurrence detected on follow-up imaging (CT or FDG-PET/CT) that is located within the SBRT target volume.
Time Frame: Up to 24 months
Population: Patients that received study treatment per protocol and were evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 49
percentage of participants | 49.69 [31.98 to 67.43]

7. Primary Outcome: Distant Metastasis-free Survival (DMFS)
Description: Percentage of patients without distant disease metastasis (progression of disease beyond local target lesion).
Time Frame: Up to 24 months
Population: Patients that received study treatment per protocol and were evaluable for response.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 49
percentage of participants | 21 [12 to NA] — Upper bound not reached.

8. Secondary Outcome: Acute Toxicities Associated With SBRT
Description: Percentage of patients that experienced acute toxicity (defined as toxicity occurring within 3 months of completion of SBRT). Toxicities were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v 4.
Time Frame: Up to 24 months
Population: Patients that received study treatment per protocol and experienced acute grade 3 þ radiation toxicity.
Measure: Number; unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 49
percentage of participants | 4.1

9. Secondary Outcome: Late Toxicities Associated With SBRT
Description: Percentage of patients that experienced late toxicity (defined as toxicity occurring after 3 months of completion of SBRT). Toxicities were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v 4.
Time Frame: Up to 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 49
percentage of participants | 0

10. Secondary Outcome: 2-year Progression-free Survival (PFS)
Description: Percentage of patients that did not experience disease progression at 2 years. For patients that undergo surgical resection, local progression will be defined as disease recurrence detected on follow-up imaging (CT or FDG-PET/CT) that is located within the SBRT target volume.
Time Frame: Up to 24 months
Population: Patients that received study treatment per protocol and were evaluable for response.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 49
percentage of participants | 32.79 [17.49 to 50.25]

11. Secondary Outcome: Time to Progression (TTP)
Description: The time from enrollment to disease progression. For patients that undergo surgical resection, local progression will be defined as disease recurrence detected on follow-up imaging (CT or FDG-PET/CT) that is located within the SBRT target volume.
Time Frame: Up to 24 months
Population: Patients that received study treatment per protocol and were evaluable for response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 49
months | 12 [7 to 27]

12. Secondary Outcome: Overall Survival (OS)
Description: The length of time from enrollment to confirmed death from any cause.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 50
months | 18 [13 to 20]

13. Secondary Outcome: Overall Survival (OS) at 1-year
Description: Percentage of patients alive at 1-year (death from any cause).
Time Frame: Up to 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 50
percentage of participants | 68

14. Secondary Outcome: Overall Survival (OS) at 2-years
Description: Percentage of patients alive at 2-years (death from any cause).
Time Frame: Up to 12 months
Population: Participants enrolled in study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 50
percentage of participants | 39.95 [24.44 to 56.68]

15. Secondary Outcome: Quality of Life (QoL) FACT-G
Description: The FACT-G is a 27 item questionnaire that assesses physical, social/family, emotional, and functional well-being, provided to patients and self-administered prior to SBRT, after completion of SBRT, and at each follow-up. The survey takes 5 minutes to complete and employs as five-point scale from 0 (not at all) to 4 (very much). Subscale scores added to obtain total score. Scoring range is between 0-108 points. Negatively worded items are reverse scored prior to summing so that higher subscale and total scores indicate better QoL.
Time Frame: Up to 24 months (before treatment (baseline), shortly after neo-adjuvant treatment, shortly after surgery, shortly after SBRT, shortly after Adjuvant treatment)
Population: Patients that completed FACT-G Quality of Life surveys.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Stereotactic Body Radiotherapy
Number analyzed (Participants) | 22
score on a scale
  Physical well-being (PWB) - Before treatment (baseline) | 24 [12 to 27]
  Physical well-being (PWB) - Shortly after neo-adjuvant treatment | 25 [23 to 27]
  Physical well-being (PWB) - Shortly after surgery | 24 [21 to 25]
  Physical well-being (PWB) - Shortly after SBRT | 23 [15 to 27]
  Physical well-being (PWB) - Shortly after adjuvant treatment | 18 [9 to 26]
  Social/family well-being (SWB) - Before treatment (baseline) | 26 [19 to 28]
  Social/family well-being (SWB) - Shortly after neo-adjuvant treatment | 28 [28 to 28]
  Social/family well-being (SWB) - Shortly after surgery | 25 [23 to 28]
  Social/family well-being (SWB) - Shortly after SBRT | 26 [20 to 28]
  Social/family well-being (SWB) - Shortly after adjuvant treatment | 17 [15 to 18]
  Emotional well-being (EWB) - Before treatment (baseline) | 17 [16 to 19]
  Emotional well-being (EWB) - Shortly after neo-adjuvant | 22 [20 to 23]
  Emotional well-being (EWB) -Shortly after surgery | 20 [16 to 22]
  Emotional well-being (EWB) -Shortly after SBRT | 21 [17 to 22]
  Emotional well-being (EWB) - Shortly after adjuvant treatment | 14 [12 to 16]
  Functional well-being (FWB) - Before treatment (baseline) | 14 [5 to 23]
  Functional well-being (FWB) - Shortly after neo-adjuvant | 20 [11 to 28]
  Functional well-being -Shortly after surgery | 22 [14 to 27]
  Functional well-being (FWB) Shortly after SBRT | 13 [11 to 21]
  Functional well-being (FWB) Shortly after adjuvant treatment | 17 [13 to 20]
  Total score - Before treatment (baseline) | 83 [52 to 95]
  Total score - Shortly after neo-adjuvant | 94 [82 to 106]
  Total score - Shortly after surgery | 85 [77 to 94]
  Total score - Shortly after SBRT | 78 [73 to 89]
  Total score - Shortly after adjuvant treatment | 64 [53 to 76]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected were collected for patients up to 24 month after initiation of treatment. All-Cause Mortality monitored for up to 48 months.
Description: Adverse Events described per NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Arm/Group | Stereotactic Body Radiotherapy
All-Cause Mortality (participants affected / at risk) | 25/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 23/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Body Radiotherapy (N=49)
Abd drain (Gastrointestinal disorders) | 1
Abdom pain (Gastrointestinal disorders) | 3
Abx diarrhea (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Delayed gastric emptying (Gastrointestinal disorders) | 2
Delirium. (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 8
Fever (General disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1
GI bleed (Gastrointestinal disorders) | 1
Hepatic bleeding (Gastrointestinal disorders) | 1
Hair thinning (Skin and subcutaneous tissue disorders) | 1
Hand foot syndrome (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 1
HHNK (Metabolism and nutrition disorders) | 1
Hyperglycemia (grade 3) (Metabolism and nutrition disorders) | 1
Leukopenia (Investigations) | 1
Lip herpetic lesion (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neuropathy (Nervous system disorders) | 1
Neutronic fever (General disorders) | 1
Neutropenia (Investigations) | 2
NG tube (Gastrointestinal disorders) | 1
Obstruction (grade 3) (Gastrointestinal disorders) | 1
Pancreatic leak (Hepatobiliary disorders) | 1
PE (Cardiac disorders) | 1
Peripheral neuropathy (Nervous system disorders) | 1
PNA (Respiratory, thoracic and mediastinal disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Right sided weakness, (Musculoskeletal and connective tissue disorders) | 1
Skin (Skin and subcutaneous tissue disorders) | 1
SMA pseudoaneurysm (Nervous system disorders) | 1
SMA pseudocyst (Hepatobiliary disorders) | 1
SMA pseuoanuersym (Nervous system disorders) | 1
SMV thrombus (Vascular disorders) | 1
Strep viridans bacteremia (Infections and infestations) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombotypenia (Blood and lymphatic system disorders) | 1
Upper GI leak (Gastrointestinal disorders) | 1
UTI (Infections and infestations) | 2
Volume depletion (Metabolism and nutrition disorders) | 1
Weight loss (Investigations) | 2
Xerstomia (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-06-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT01357525/Prot_SAP_000.pdf